CLINICAL TRIAL: NCT01625910
Title: For the Health of Our Children--Clinic Based Treatment of Childhood Obesity: The Feasibility of Recruitment and the Effectiveness of a Low-intensity Stage
Brief Title: For the Health of Our Children--Clinic Based Treatment of Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1107M02462
Record Dates: First submitted 2012-04-10; First posted 2012-06-22 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Obesity
Keywords: Childhood obesity treatment; Motivational interviewing
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- behavioral counseling (Experimental): Receive counseling via motivational interviewing seeking to encourage health eating habits and increased physical activity
  Interventions: Behavioral: Behavioral counseling
- Instructions in school readiness and performance (Placebo Comparator): Parents receive instructions in school readiness and performance
  Interventions: Behavioral: Behavioral counseling

INTERVENTIONS:
Behavioral: Behavioral counseling — Counseling of parents to improve their child's diet and physical activity
  Other Names: Motivational Interviewing; Pediatric obesity treatment

SUMMARY:
Childhood obesity is a major public health problem in the U.S. Currently approximately one in three children is considered overweight or obese. Most overweight children grow to become overweight adults. It is unclear how effective pediatricians and other primary care physicians can be in assisting overweight children to normalize their body weight. Expert guidelines have been established, but are currently untested.

This study will randomize overweight and obese children between the ages of 4 and 8 years old to either the recommended treatment guidelines or a control (non-intervention) group.

The purpose of this study is to evaluate the ability (a) to recruit overweight children between the ages of 4 and 8 years old (b) to remeasure the children three months after enrollment and (c) to reduce childhood obesity via implementation of the recommended treatment guidelines.

DETAILED DESCRIPTION:
3. Research Plan:

a. Specific Aims and Hypothesis: In 2007, an expert committee, composed of representatives from 16 major clinical organizations (including the PI of this proposal), published recommendations for primary care office-based treatment of childhood obesity. Seeking both clinical and cost-effectiveness, the recommendations call for staged treatment that starts with low intensity, and then, if unsuccessful, increases to a higher frequency of visits. The committee acknowledged that this staged approach "has not been evaluated." Recent reviews conclude that treatment of childhood obesity can be efficacious. However, most studies were conducted in highly controlled tertiary care research settings and involved a large number of direct contact hours (e.g. many with ≥ 35 contact hours). Research evaluating the translation of these encouraging findings into more real-world clinical settings has been lacking. Specifically, there is little research assessing (1) the feasibility of recruitment from primary care clinics or (2) whether low intensity treatment (i.e. the initial phase of the staged approach recommended by the expert committee) has any benefit on weight loss.

* Aim #1: To assess the feasibility of recruiting overweight and obese children, ages 4-8 years, from a large, urban pediatric primary care clinic, randomizing them to either low-intensity treatment or a control group, and then re-measuring them at approximately 3-months from the date of recruitment.

  o Our hypothesis is that we will be able to recruit approximately 70 parent/child dyads and re-measure 80% at 3-months.
* Aim #2: To evaluate whether the proportion of children who decrease their BMI z-score over a 3-month period is higher in those randomly assigned to the intervention group compared with those in the control group.

  * Our hypothesis is that the intervention will result in a larger proportion of children decreasing BMI z-score over a 3-month period.

Results from Aims 1 and 2 will be used to plan for an NIH proposal. If the low intensity treatment of this proposal shows a trend toward improvement over usual care, this will justify a full scale, R01 trial testing the complete recommendations of the expert committee. If few subjects in the intervention group have decreasing BMI z-scores, then a smaller NIH trial would be needed to test an amended low-intensity treatment stage with more parent/child contact (e.g. emails, home visits, phone calls).

ELIGIBILITY:
Inclusion Criteria:

* any patient at the participating clinic between the ages of 4-8 years who have a BMI ≥ the 85th percentile

Exclusion Criteria:

* emergent health concern
* serious chronic health concern or recent gastrointestinal illness which may have resulted in weight loss
* on medications known to affect weight

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Stovitz, MD, MS, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Fairview Children's Clinic, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment occurred from Sept 2011 - May 2012. Permission was first obtained from the clinicians and then the parent-child dyads who agreed gave written parental consent and, if the child was at least 8 years of age, child assent. Prior to randomization, a parent answered the intake survey and child ht and wt were re-measured by the RA.
Pre-assignment Details: After enrollment, the children were randomly assigned to either the intervention or control group. The intervention and control group protocols began on the day of enrollment, immediately after group assignment
Groups:
- Intervention - Behavioral Counseling: The intervention group received management patterned after the
- Control: On the day of enrollment, after randomization to the control/usual care group, the RA provided age- and ability-appropriate informational hand-outs on school readiness and/or performance.
Period: Overall Study
Arm/Group | Intervention - Behavioral Counseling | Control
Started | 35 | 37
Completed | 32 | 33
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: Random allocation resulted in 35 participants in the intervention group and 37 in the control group. However, one participant in the control group was not included in the final analyses due to an interim injury (unrelated to the study) and prolonged cast treatment.
Groups:
- Intervention - Behavioral Counseling: The intervention group received management patterned after the "Prevention plus, Stage 1" treatment recommended by the expert panel and approved by the committee. Counseling was primarily directed toward the parents. The RA used motivational interviewing (MI) techniques as an entry way to discuss healthy lifestyle habits around eating and physical activity (e.g., open-ended questions, reflective listening, discrepancy questions, eliciting change talk). Evidence-based recommendations for childhood obesity treatment were discussed with the parent; such as, eating breakfast daily, eating ≥ 5 servings of fruits and vegetables/day, avoidance of skipping meals, watching ≤ 2 hours of screen time/day, minimizing or eliminating sugar-sweetened beverages, encouraging family meals at home, and being physically active ≥ 1 hour/day.
  There were monthly follow-up phone calls to try and encourage continued success in healthy lifestyle choices.
- Total: Total of all reporting groups
Arm/Group | Intervention - Behavioral Counseling | Control | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 37 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 16 | 19 | 35
BMI- Z score [Mean (Standard Deviation); unit: z-score units] — At baseline and the 3-month follow up visit, the children's heights and weights were measured by trained RAs. The measurements at follow-up were done by an RA, blinded to group assignment. Height and weight were measured with the child in light indoor clothing, with shoes and socks removed. RAs measured height (cm), in triplicate, using a Shorr height board, and reported the mean of the three readings. Weight was measured using a Tanita scale. Age- and gender-specific BMI Z-scores were calculated using the US CDC 2000 growth charts.
  z-score units | 1.90 (0.55) | 1.89 (0.82) | 1.90 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index Z-score Change
Description: Change in body mass index z-score change over the three month time period
Time Frame: Three months
Population: All enrolled were analyzed with one exception (due to injury and prolonged cast treatment). An intent-to-treat analysis required that, for those who did not have the follow-up measurement, data were filled in using the experience of those in the control group who had follow-up measurements.
Measure: Mean (Standard Error); unit: BMI z-score change
Arm/Group | Intervention - Behavioral Counseling | Control
Number analyzed (Participants) | 35 | 36
BMI z-score change | -0.02 (0.05) | -0.08 (0.05)
Statistical Analysis 1: Comparison: Intervention - Behavioral Counseling vs Control; Baseline data by group assignment status (intervention or control) using means of the calculated BMI z-scores (U.S. CDC-2000 growth charts) implemented by applying the published LMS (shape, median, and scale) age- and sex/gender-specific parameters. Because of random assignment of a reasonably large number of children, an unadjusted analysis of change in outcomes between intervention and control groups is presented as well as the covariate-adjusted analysis of differences in changes; Test type: Superiority or Other; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.10 to 0.21], Standard Error of Mean 0.05

2. Secondary Outcome: Sugar Sweetened Beverages
Description: Change in reported intake of sugar sweetened beverages
Time Frame: Three months
Population: Intention to treat analysis
Measure: Mean (Standard Error); unit: cans per day
Groups:
- Intervention Group: The survey done at baseline and follow-up asked about daily cans of sugar-sweetened beverages.
  Estimate is for Change in cans of sugar sweetened beverages per day
- Control: Change in cans of sugar sweetened beverages per day
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 35 | 36
cans per day | -0.14 (0.20) | 0.03 (0.20)
Statistical Analysis 1: Comparison: Intervention Group vs Control; unadjusted net difference between groups; Test type: Superiority or Other; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.74 to 0.40], Standard Error of Mean 0.20

ADVERSE EVENTS:
Arm/Group | Intervention - Behavioral Counseling | Control
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

LIMITATIONS AND CAVEATS:
There were no adverse events during this 3-month trial comparing a parent-based behavioral intervention with usual care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes